CLINICAL TRIAL: NCT05484986
Title: Relationship Between Nursing Students' Personality Traits and Competence in Workplace Violence Management in Turkey: A Cross-sectional Study
Brief Title: Nursing Students' Personality Traits and Competence in Workplace Violence Management
Status: Completed | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Derya Akça Doğan, Research Assistant, Uludag University
Other Study IDs: DDogan
Record Dates: First submitted 2022-07-28; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Exposure to Violent Event; Nursing Student; Personality; Violence; Workplace Bullying
Keywords: exposure to violence; nursing student; personality; violence; workplace
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nursing students
  Interventions: Other: A questionnaire with 47 items

INTERVENTIONS:
Other: A questionnaire with 47 items — A form consisted of questions on introductory characteristics (age, sex, and class, among others), Big Five Inventory (BFI) to evaluate personality traits, and Management of Workplace Violence Competence Scale for Nursing Students in Areas of Clinical Practice.

SUMMARY:
Aim: The aim of this study was to determine the relationship between nursing students' personality traits and competence in workplace violence management.

Background: Violence against nursing students is a growing concern in nursing education, clinical practice, and professional development and needs to be managed.

Design: A cross-sectional study. Methods: This study was conducted with 321 nursing students in the summer of 2022.

ELIGIBILITY:
Inclusion Criteria:

* Being in the nursing students at the research university,
* Being in the >18 years age,
* Agree to participate in the study

Exclusion Criteria:

* Being in the <18 years age,
* Disagree to participate in the study

Age Groups: Child, Adult, Older Adult
Study Population: Nursing students
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2022-05-14 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
To determine nursing students' personality traits | 1 month
  İn this study personality traits of nursing students was examined using the Big Five Inventory (BFI), and management of workplace Vvolence competence of nursing students was examined using the Management of Workplace Violence Competence Scale for Nursing Students in Areas of Clinical Practice.
To determine nursing students' competence in workplace violence management | 1 month
To determine the relationship between nursing students' personality traits and competence in workplace violence management | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No